CLINICAL TRIAL: NCT06608745
Title: CAS vs Tecnica Chirurgica Standard Nella Protesi Totale di Ginocchio: Confronto Dei Risultati Clinico-funzionali
Brief Title: CAS vs Standard Technique in TKA: Comparison of Clinical and Functional Results
Acronym: CAS-K
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CE-AVEC 572/2023/Sper/IOR
Record Dates: First submitted 2024-09-10; First posted 2024-09-23 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Knee Arthroplasty, Total

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- conventional total knee arthroplasty surgery (Active Comparator)
  Interventions: Procedure: conventional total knee arthroplasty
- computer-assisted total knee arthroplasty surgery (Experimental)
  Interventions: Procedure: computer-assisted total knee arthroplasty

INTERVENTIONS:
Procedure: conventional total knee arthroplasty — total knee arthroplasty performed with conventional technique
  Arms: conventional total knee arthroplasty surgery
Procedure: computer-assisted total knee arthroplasty — total knee arthroplasty performed with imageless computer-assisted surgery
  Arms: computer-assisted total knee arthroplasty surgery

SUMMARY:
The study involves the enrollment of a sample of patients with indication for total knee replacement surgery in order to compare the conventional surgical technique currently used in the reference departments with the surgical technique with the aid of computer-assisted navigation.

The comparison between the two techniques will be performed in terms of clinical-functional results, perioperative bleeding and healthcare costs (surgical time, hospital stay).

The research protocol involves the participation of 160 total patients divided into two groups, of 80 patients each, by type of surgical technique.

ELIGIBILITY:
Inclusion Criteria:

* Patients with primary or secondary gonarthrosis with indication for knee arthroplasty with primary implant
* Males and females aged ≥ 45
* Willingness to participate in the study
* Acquisition of informed consent to participate

Exclusion Criteria:

* Patients who are not capable of understanding and willing, and therefore unable to express consent to participation in the study
* Patient refusal to participate in the study and to sign the informed consent
* Nickel allergy (suspected or diagnosed)
* Pregnant women or women of childbearing age who cannot exclude pregnancy

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2024-02-12 (Actual); Primary Completion 2026-08-12 (Estimated); Study Completion 2026-08-12 (Estimated)

PRIMARY OUTCOMES:
Knee Society Score (KSS) | From enrollment to 12 months post-operative followup
  Knee Society Clinical Rating System (KSS):
  there are 2 section, "Knee Score" section and a "Functional Score" section; both sections are scored from 0 to 100 with lower scores being indicative of worse knee conditions and higher scores being indicative of better knee conditions
Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | from enrollment to 12 months post-operative followup
  Set of standardized questionnaires used by health professionals to evaluate the condition of patients with osteoarthritis of the knee and hip, including pain, stiffness, and physical functioning of the joints.
  The score measures five items for pain (score range 0-20), two for stiffness (score range 0-8), and 17 for functional limitation (score range 0-68).
  Higher scores indicate worse pain, stiffness, and functional limitations.
NRS scale | from enrollment to 12 months post-operative followup
  Numeric Pain Rating scale is a unidimensional measure of pain in which a patient selects a whole number (0-10 integers) that best reflects the intensity of his/her pain.
  0 = no pain, 10 = worst pain possible

SECONDARY OUTCOMES:
surgical time | the day of surgical procedure
complications | from surgery to 12 month follow-up
  using Clavien Dindo classification of surgical complications
delta hemoglobin | from surgery to discharge, up to 4 weeks
  For each patient blood loss will be assessed by measuring the difference in hemoglobin (g/dL) on the preoperative blood sample VS last blood sample before discharge
Transfusions | from surgery to discharge, up to 4 weeks
  It will be accounted the number of blood transfusions that patients may need during the hospital stay until discharge
hospital stay | from surgery to discharge, up to 4 weeks
  days of hospital stay from surgery to discharge

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Ortopedico Rizzoli, Bologna, Italy